CLINICAL TRIAL: NCT00396669
Title: A Brain Imaging Study Into Nicotine Induced Dopamine Release in Cigarette Smokers, Using 11 C Raclopride in Positron Emission Tomography (PET)
Brief Title: A Brain Imaging Study Into Nicotine Induced Dopamine Release in Cigarette Smokers.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, VEINSHTEIN AVIV, Senior Research Fellow, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 291006 HMO-CTIL
Record Dates: First submitted 2006-11-06; First posted 2006-11-07 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Tobacco Use Disorder
Keywords: Nicotine; Dopamine; Imaging; Raclopride; Addiction; Genetics
MeSH Terms: conditions — Tobacco Use Disorder; Behavior, Addictive | interventions — Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dopamine release (Experimental)
  Interventions: Drug: Bupropion

INTERVENTIONS:
Drug: Bupropion — We measure dopamine release at the striatum using 11 C Raclopride at baseline and after smoking a cigarette
Drug: Bupropion — Brain imaging after treatment with Bupropion
  Other Names: Zyban

SUMMARY:
Dopamine (DA) plays a critical role in nicotine (and other) addiction and this drug is known to release DA in brain areas mediating reward and motivational processes. Although imaging studies show that release of DA follows smoking, little is known regarding how common genetic polymorphisms for three genes associated in some studies with smoking (dopamine D2 receptor, dopamine and serotonin transporter) interact with smoking status and modulate individual differences in nicotine-induced DA release and dopamine receptor occupancy, in vivo. The current proposal combines brain imaging and genomics ('imaging genomics') towards partially unraveling the complex relationship between smoking phenotype and common polymorphisms. Understanding whether genetic factors contribute to inter-individual variability in smoking is crucial for interpreting imaging results in the context of disease pathology. We hypothesize that a model of vulnerability to addiction based on interactions between genotype, receptor and transporter availability and in vivo nicotine-induced DA release will elucidate some of the fundamental neurochemical and neurogenetic circuits underlying addiction.

DETAILED DESCRIPTION:
Dopamine plays a critical role in nicotine(and other) addiction and this drug is known to release DA in brain areas mediating reward and motivational processes. Although imaging studies show that release of DA follows smoking, little is known regarding how common some genetic polymorphisms proposed to play a role in nicotine dependence (e.g. DRD2, DAT and the serotonin transporter or SERT) interact with smoking status (non-smoker, ex-smoker, light smoker, present smoker) and modulate individual differences in nicotine-induced DA release and dopamine receptor occupancy, in vivo. Individual differences in dopaminergic tone could result in an under-stimulation of reward circuits which could put subjects at greater risk for seeking drug stimulation (that releases DA) as a means to compensate for this deficit and to temporarily activate these reward circuits. The current proposal combines brain imaging and genomics towards unraveling the complex relationship between smoking phenotype and common polymorphisms. Understanding whether genetic factors contribute to inter-individual variability is crucial for interpreting imaging results in the context of disease pathology.

Nicotine dependence is a complex process including initiation of smoking, persistence and difficulty in quitting. By comparing receptor occupancy, nicotine-induced DA release, and common genetic polymorphisms across smoking behaviors we will better understand the complex interactions between genetic makeup, personality and the several stages of nicotine addiction.

ELIGIBILITY:
Inclusion Criteria:

* smokers who smoked 15 cigarettes/day and who met the DSM-IV criteria for nicotine dependence

Exclusion Criteria:

* Subjects who are diagnosed as suffering from psychotic illness according to DSM-IV (Axis 1)22, or with a history of CNS disease, a history of infection that might affect CNS (HIV, syphilis, cytomegalovirus, herpes), or a history of head injury with loss of consciousness will be excluded.

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2007-07; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Dopamine D2 receptor occupancy before and after smoking a cigarette with nicotine | 30 minutes

SECONDARY OUTCOMES:
Subjective measures of craving, anxiety and depression. | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Aviv M Weinstein, Ph.D, Principal Investigator — Hadassah Medical Organization; Moshe Bocher, M.D, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel